CLINICAL TRIAL: NCT00899080
Title: Screening of Cathepsin G Levels in Multiple Myeloma Patients Receiving Treatment With Thalidomide/Lenalidomide Within the ECOG Trials E1A00 and E4A03
Brief Title: Studying Blood Samples From Patients With Multiple Myeloma Who Were Treated With Thalidomide or Lenalidomide
Status: Completed | Type: Observational
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CDR0000600320; ECOG-E4A03T2
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2017-05-17 (Actual); Status verified 2017-05

CONDITIONS: Multiple Myeloma and Plasma Cell Neoplasm
Keywords: stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Gene Expression Profiling; Reverse Transcriptase Polymerase Chain Reaction; Immunoenzyme Techniques; Platelet Aggregation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective

INTERVENTIONS:
Genetic: gene expression analysis
Genetic: reverse transcriptase-polymerase chain reaction
Other: immunoenzyme technique
Other: laboratory biomarker analysis
Other: platelet aggregation test

SUMMARY:
RATIONALE: Studying samples of blood from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer. It may also help doctors predict how patients will respond to treatment.

PURPOSE: This research study is looking at blood samples from patients with multiple myeloma who were treated with thalidomide or lenalidomide.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To analyze the mechanism of development of thalidomide/lenalidomide-induced venous thromboembolism (VTE) in patients with multiple myeloma treated on clinical trial ECOG-E4A03 or E-E1A00.
* To determine the intensity, dynamics, and specificity of cathepsin G (CG) upregulation in response to thalidomide and lenalidomide treatment.
* To determine the specificity and threshold levels of CG for induction of platelet aggregation in response to thalidomide and lenalidomide and the resulting risk for VTE development.

OUTLINE: Blood samples obtained before, during, and after treatment with thalidomide or lenalidomide from patients previously enrolled on clinical trial ECOG-E4A03 or E-E1A00 are analyzed to determine the total content of cathepsin G (CG) via ELISA; to determine mRNA levels of CG via RT-PCR; and for platelet aggregation studies. Blood samples are collected from healthy volunteers for platelet preparation.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Meets 1 of the following criteria:

  * Diagnosed with multiple myeloma and treated with thalidomide or lenalidomide on clinical trial ECOG-E4A03 or E-E1A00
  * Healthy volunteer

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Max Age: 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Samples submitted for research from patients enrolled on E4A03 or E1A00
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2008-07-04 (Actual); Primary Completion 2008-08-04 (Actual); Study Completion 2008-08-04 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with failed disease based on expectations for changes in cathepsin G (CG) levels | 1 month

SECONDARY OUTCOMES:
Mechanism of development of thalidomide/lenalidomide-induced venous thromboembolism (VTE) | 1 month
Intensity, dynamics, and specificity of CG upregulation in response to thalidomide and lenalidomide treatment | 1 month
Specificity and threshold levels of CG for induction of platelet aggregation in response to thalidomide and lenalidomide and the resulting risk for VTE development | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Lentzsch, MD, PhD, Study Chair — University of Pittsburgh